CLINICAL TRIAL: NCT01797640
Title: Intramedullary Nailing of Tibia Fractures in the Presence of Medial or Posterior Malleolar Fractures
Brief Title: Intramedullary Nailing of Tibia Fractures
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Eric Kubiak, M.D., University of Utah
Other Study IDs: 50553
Record Dates: First submitted 2013-01-04; First posted 2013-02-22 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Tibial Fractures; Malleolar Fractures
Keywords: Tibia Fractures; Medial Fractures; Posterior Malleolar Fractures
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Currently, the treatment of choice for tibial fracture is intramedullary nailing. This procedure has been shown to have low rates of infection, high rates of bone healing, and a faster return to weight bearing and activity in comparison to conservative treatment. In concurrent fractures of the posterior or medial malleolus and the tibia, it is now common to identify, reduce, and fix the malleolar fracture prior to intramedullary nailing of the tibia. In this retrospective study, our aim is to establish that reducing malleolar fractures prior to tibial nailing is a safe treatment in which the reduction of the malleolus is maintained intraoperatively, postoperatively, and remains reduced until the fracture has healed.

ELIGIBILITY:
Inclusion Criteria:

* All patients, 18+ years of age, that have been treated at the University of Utah over the past five years for tibial fracture combined with medial or posterior malleolar fracture.

Exclusion Criteria:

* None

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prospectively evaluating all patients that have been treated at the University of Utah over the past five years for Tibial Fracture combined with medial or posterior malleloar fracture.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2012-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Malleolar involvement in tibial fracture | 6 Week Post-Op
  Currently the treatment of choice for tibial fracture is intramedullary nailing. This procedure has been shown to have low rates of infection, high rates of bone healing, and a faster return to weight bearing and activity in comparison to conservative treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Kubiak, Principal Investigator — Orthopedic Surgery Operations
Locations (1):
- University of Utah Orthopedics Center, Salt Lake City, Utah, United States